CLINICAL TRIAL: NCT04377685
Title: Prediction of Clinical Course in COVID19 Patients Using Unsupervised Classification Approaches of Clinical, Biological and the Multiparametric Signature of the Chest CT Scan Performed at Admission
Brief Title: Prediction of Clinical Course in COVID19 Patients
Acronym: COVID-CTPRED
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: INSA Rennes (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre National pour le Recherche Scientifique (CNRS) (Unknown); Université de Lyon (Unknown); Jean Monnet University (Other)
Responsible Party: Sponsor
Other Study IDs: 20CH109; IRBN652020/CHUSTE (Other: Comité d'éthique du CHU de Saint-Etienne)
Record Dates: First submitted 2020-05-05; First posted 2020-05-06 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: COVID 19
Keywords: COVID 19; chest CT scan
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID19 patients: Patient tested positive for SARS-CoV-2 who had a CT scan
  Interventions: Other: CT-Scan

INTERVENTIONS:
Other: CT-Scan — Chest CT scan on admission to the hospital

SUMMARY:
In the context of the COVID19 pandemic and containment, chest CT is currently frequently performed on admission, looking for suggestive signs and basic abnormalities of COVID19 compatible viral pneumonitis pending confirmation of identification of viral RNA by reverse-transcription polymerase chain reaction(PCR), with a reported sensitivity of 56-88% in the first few days, slightly higher than PCR (60%) (1). Nevertheless, currently established radiological abnormalities are not specific for COVID19 and the specificity of the chest CT is ~25% when PCR is used as a reference (1). Deconfinement and its consequences will complicate the triage of COVID patients and the role of the scanner, with the expected impact of a decrease in the prevalence of infection in the emergency department and an increase in the number of "all-round" patients, including patients with non-COVID viral infiltrates or pneumopathies.

In addition, there are currently no imaging criteria to complement the clinical and biological data that can predict the progression of lung disease from the initial data.

DETAILED DESCRIPTION:
In image processing, computational medical imaging has demonstrated its ability to predict a therapeutic response or a particular evolution after extracting relevant anatomical, functional or even non-visually perceptible information from the volume of images, making it possible to construct a powerful radiomic signature or to use robust anatomical/functional measurements to provide estimates of ventilation or vascular state. By combining these data extracted from the scanner with the standard clinical-biological data produced at admission during triage, our ambition is to build a predictive model using unsupervised classification approaches capable of helping predict clinical evolution with the aim of optimizing the management of the resource.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* clinical suspicion of COVID-19 confirmed by RT-PCR
* CT scan at ER admission
* RT-PCR sampling

Exclusion Criteria:

* CT scan failure or loss of CT data
* RT-PCR initial results unavailable

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient admitted to the emergency room of COVID-19 confirmed by RT-PCR
Sampling Method: Non-Probability Sample
Enrollment: 826 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2020-12-26 (Actual)

PRIMARY OUTCOMES:
diagnostic of COVID disease composite | On admission to the hospital
  The diagnostoc of COVID disease is composite of:
  * CT features wich will include presence/location/laterality of morphological CT abonormal densities (ground glass opacities, consolidations, reticulations),
  * pulmonary vessels size,
  * distribution and abnormalities,
  * local / global CT-ventilation index (CT-VI) severity,
  * radiomic features (shape features, 1st-order and 2nd order statistics)
  Analysis of CT-Scan results.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre CROISILLE, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No